Official Title: Weight Management for Adults with Mobility Related Disabilities

NCT Number: 04046471

Approval Date: January 26, 2024

Document: Study Protocol with Statistical Analysis Plan

### **AIMS AND HYPOTHESES**

Individuals with mobility related disabilities (MRDs) represent a sizeable and growing segment of the U.S. adult population, with high rates of obesity, and limited options for successful weight management. Obesity in adults with MRDs increases the risk of chronic disease, and may limit the ability to ambulate, either with or without assistive devices (wheelchair, cane etc.), perform transfers (wheelchair users), increase the risk for pressure sores, respiratory problems, carpal tunnel syndrome, and interfere with self-care, and reduce participation in daily activities. Adults with MRDs face numerous barriers to participation in traditional weight management programs including the lack of affordable, accessible transportation to attend on-site meetings or engage in physical activity (PA), lack of accessible recreational facilities with accessible fitness equipment, and difficulty with food shopping and meal preparation. The 2005 Surgeon General's Call to Action to Improve the Health and Wellness of Persons with Disabilities, and numerous subsequent government sponsored reports, have highlighted the need for accessible health promotion efforts to reduce health disparities between adults with and without MRDs. However, a limited number of intervention strategies, specific to weight management in adults with MRDs. have been developed and evaluated. As described in this proposal, our group has evaluated an enhanced version of the Stop Light Diet (eSLD = SLD+portion-controlled meals and low calorie shakes) for weight management in a sample of 126 adults with MRDs. The eSLD simplifies meal planning, food shopping and meal preparation. When prescribed in conjunction with a monthly behavioral intervention, delivered in an individual home visit format, the eSLD resulted in significantly greater weight loss when compared with a conventional meal plan diet at 6 mos. (eSLD = -4.1%, meal plan = -2.3%, p=0.02) and 12 mos. (eSLD = -6.2%, meal plan = -0.6%, meal plan = -0.6%)p=0.005). Although these results are encouraging, alternative strategies to improve outcomes and to deliver weight management to larger numbers of adults with MRDs in a cost-effective manner, are warranted. Thus, the proposed two-arm randomized trial will compare weight loss (6 mos.) and maintenance (18 mos.) between an individual home visit intervention (IH), using an enhanced version of the protocol used in our previous trial, and an intervention delivered remotely via video conferencing to groups of overweight/obese adults with MRDs in their homes (GR). Both interventions will be delivered in a format that eliminates the transportation barrier, prescribed an eSLD, and will self-monitor body weight using electronic scales. The GR arm will include group behavioral counseling and group PA delivered remotely via video conferencing (Zoom<sup>TM</sup> software) on a tablet computer (iPad mini) to participants in their homes, and use commercially available web-based applications for self-monitoring/participant feedback for diet (Lose It! software) and PA (Fitbit activity tracker). This approach reduces barriers to both behavioral session attendance and PA, provides timely feedback relative to diet and PA, and promotes interaction and support in a group who are often socially isolated. The IH arm, which represents a modified version of the protocol used in our previous trial, will include behavioral counseling delivered during individual home visits, a prescription for self-directed PA, and selfmonitoring of diet and PA using conventional paper and pencil self-reports. Both groups will receive identical attention with 2 interventions having the potential for clinically meaningful weight loss, i.e., ≥ 5%. This trial will address the following primary, secondary and exploratory aims.

**Primary aim:** <u>To compare mean weight loss between the GR and IH arms across 6 mos.</u> We expect significantly greater weight loss in the *GR* compared to the *IH* arm.

**Secondary aims.** To compare the GR and IH arms on the following: 1) Mean weight loss (0-18 mos.); 2) The proportion of participants who achieve clinically significant weight loss ( $\geq$  5% from baseline) at 18 mos.; 3) Changes in cardiovascular disease risk factors (blood pressure, total, HDL and LDL cholesterol, triglycerides, HbA1c for diabetics, waist circumference) from 0-6 and 0-18 mos.; 4) Changes in quality of life from 0-6 and 0-18 mos. We expect more favorable changes in all secondary outcomes in the GR compared with the IH arms. 5) Cost and contingent valuation analysis to compare costs between the GR and IH arms. Based on our experience with remote delivery for weight management using both group phone (DK76063) and virtual reality formats (DK94833), we expect GR to be less expensive than the IH arm.

**Exploratory aims.** *Initial weight loss is highly predictive of longer-term weight loss; therefore, we will examine the influence of the following variables on weight loss at 6 and 18 mos.*: behavioral session attendance, compliance with the recommendations for diet (energy intake, number of meals /shakes, servings of fruits/vegetables), PA (min of moderate-vigorous PA, min sedentary time), and self-monitoring of diet and PA, self-efficacy for dietary change and PA, dietary self-regulation, social support for diet/PA, barriers to PA, sleep, and medications.

# **BACKGROUND/SIGNIFICANCE**

Mobility related disabilities (MRDs)-Prevalence/descriptive characteristics. MRDs are the most frequently reported type of disability in U.S. adults (1-6). The estimated prevalence of MRDs in the U.S. varies across surveys due to differences in sampling strategies, definitions of disability, and age ranges reported (7). For example, data from the 2013 Behavioral Risk Factor Surveillance System (BRFSS) indicated the prevalence of MRD was 13% in individuals ≥18 yrs. (1), while the prevalence of mobility limitations in the same age group was 6.1% in the 2011-2014 National Health Interview Survey (NHIS) (3). Data from the U.S. Census Bureau's 2015 American Community Survey indicated 6.6% of adults age 18-64 yrs. reported an ambulatory disability (6), while data from the US Census Bureau Survey of Income and Program Participation (May-August 2010) indicated 12.6% of individuals ≥ age 15 yrs. reported limitations in ambulation (2). Regardless of the variation in prevalence estimates, adults with MRDs represent a sizeable segment of the U.S. population. Increased survival rates from traumatic injuries or premature birth, increased life expectancy for both congenital and acquired disabilities, and the aging of the population, will contribute to future increases in the prevalence of MRDs. The prevalence of MRDs is higher in females, older individuals, ethnic minorities, the unemployed, and in adults with lower levels of education and annual household income (1, 7). Adults with MRDs are less likely to be physically active (8-13), more likely to have poor diet quality (14, 15), higher rates of chronic conditions (16-20), risk factors for chronic conditions (16, 21-24), and an increased risk for all-cause mortality (25, 26), compared with their non-disabled counterparts.

**Obesity prevalence/consequences**. The prevalence of obesity (BMI  $\geq$  30 kg/m²) in adults with MRDs is significantly greater than their non-disabled counterparts (6, 7, 16). However, the prevalence of obesity varies by data source, definition of MRD, and the use of self-report or measured height and weight for the calculation of BMI. Similar to non-disabled adults (27, 28), those with MRDs tend to overestimate height and underestimate weight (29) resulting in an

underestimate of obesity prevalence. Self-report data from the 2015 BRFSS survey indicated a higher prevalence of obesity in individuals with (39.9%) compared to those without disability (25.4%) (6). NHIS data indicated a higher prevalence of obesity in those reporting mobility (54.5%) compared with non-mobility limitations (34.5%) (8). The prevalence of obesity in adults with MRDs (≥ 20 yrs.) from the NHANES 1999-2010, using height and weight measured at a mobile clinic, was 50.9% (16). Similar to non-disabled adults, obesity in adults with MRDs is associated with unfavorable chronic disease risk factors (higher blood pressure, total cholesterol, glucose, CRP and lower HDL-cholesterol) (16), and contributes to higher rates of cardiovascular disease and other chronic conditions (19). The combination of MRDs and obesity may limit the ability to ambulate and perform transfers (wheelchair users) (30), increases the risk for pressure-sores (4, 31), respiratory problems (32), carpal tunnel syndrome (33), and interferes with self-care, reduces quality of life, and increases health care expenditures (34-36).

Health promotion. The 2005 Surgeon General's Call to Action to Improve the Health and Wellness of Persons with Disabilities, and subsequent reports from agencies including the Institute of Medicine (37), the National Council on Disability (38), Healthy People 2010 and 2020 (39, 40), and the Patient Protection and Affordable Care Act (2010) (41) suggest that *disability* and *health* are not mutually exclusive, and have highlighted the need for accessible health promotion efforts to prevent secondary conditions and reduce health disparities among individuals with disabilities. In response, programs addressing physical activity (PA) (42-44), healthy eating, stress management, and the development of supportive interpersonal relationships, such as Living Well with a Disability (45-47), Healthy Lifestyles for People with Disabilities (48), and others (31, 49, 50) have been implemented. These programs have reduced the prevalence of secondary conditions (51) and health care expenditures (46), increased general health behaviors (47), increased self-efficacy for a variety of life skills (49, 50), and increased PA (42, 44). However, few interventions have specifically addressed weight management, or compared the effectiveness of different weight management strategies, in adults with MRDs.

Weight management. A 2014 systematic review (52) identified 15 weight loss trials in adults with mobility-impairing neurological and musculoskeletal conditions. The majority of these trials (60%) involved older adults with osteoarthritis and reported weight loss that failed to exceed the ≥ 5% threshold defined as clinically meaningful (53). Similar results were shown in trials including ambulatory and non-ambulatory, and both younger and older individuals with MRDs. For example, Rimmer et al (54) completed a 9 mo. trial in 102 overweight/obese adults (age~47 yrs.) with MRDs (~63% non-ambulatory) randomized to 1 of 3 groups: personalized PA plan, personalized PA+nutrition plan, or non-intervention control. The nutrition plan included increased consumption of fruits, vegetables and fiber, and reduced consumption of fat, but did not specify a level of energy intake. Interventions were delivered by individual phone calls conducted by health coaches assisted by a web-based computer support system. Participants received weekly calls to develop/implement a PA or PA+nutrition plan, monitor progress, and resolve barriers. Call frequency was reduced to 2/mo. (mos. 5-7) and 1/mo. (mos. 8-9). Results from the 91 participants completing the trial indicated a small weight reduction in the PA only group (-2.4%, p<0.05), while weight was unchanged in the PA+nutrition group (-0.6%, p > 0.05), and significantly increased in controls (+3.1%, p <0.05). Chen et al. (55) evaluated a 12 wk. weight loss intervention that included an energy reduced diet, increased PA, and weekly on-site

group behavioral counseling in 16 overweight/obese adults with chronic spinal cord injury (SCI, ≥ 1 yr., age ~ 44 yrs., 100% non-ambulatory) with a 12 wk. follow-up. Results indicated small, but statistically significant weight loss at both 12 (-3.8%, p< 0.0004) and 24 wks. (-3.0%, p<0.01). Betts & Froehlich-Grobe (56) recently reported -4.8% weight loss in a 20-wk. trial in a small sample (n=10) of adults (age ~49 yrs.), with MRDs (80% non-ambulatory) using the Diabetes Prevention Group Lifestyle Balance program delivered by weekly group phone calls (1-12 wks.), with 3 additional calls over the following 8 wks. Radomski et al (57) reported a median weight loss of 5.7% in a small sample of adults (n=10, age ~ 53 yrs.) with SCI (100% non-ambulatory) following a 12 wk. exercise and education intervention consisting of individualized diet and exercise recommendations, weekly on-site group nutrition and exercise education, and twice weekly exercise sessions (both group and individual). Our group recently published results from a 12 mo. trial (6 mos. weight loss, 6 mos. maintenance, NIDRR 133G090230, M. Saunders, PI) in a sample of 126 low income (~83% unemployed), overweight/obese (BMI ~ 44 kg/m<sup>2</sup>), adults (age ~ 51 yrs.) with MRDs, 71% used wheelchair or an assistive device for walking (58). Participants were randomized to a behavioral weight loss intervention that included monthly home visits by a health educator and a reduced energy conventional meal plan, or an enhanced Stop Light Diet (eSLD; 1,200-1,500 kcal/d), selfmonitoring (logs), and optional PA. The Stop Light Diet, developed for use in children (59), categorizes foods by energy content corresponding to a traffic light, i.e., red (eat sparingly), yellow (eat moderately), and green (eat freely). We enhanced the SLD by encouraging daily consumption of 2 portion-controlled meals (≤ 300 kcal each), 2 high volume low energy shakes (100 kcal each), and ≥ five 1-cup servings of fruits/vegetables. Mean percent weight loss was significantly greater in the eSLD compared with the meal plan groups at 6 mos. (eSLD = -4.1%, meal plan = -2.3%, p = 0.024) and 12 mos. (eSLD = -6.2%, meal plan = -0.6%, p = 0.005). The percentage of randomized participants achieving ≥ 5% weight loss at 6 mos. did not differ by group (eSLD = 36%, meal plan = 23%, p = 0.15). However, the percentage of participants losing ≥ 5% of baseline weight at 12 mos. was significantly higher in the eSLD (36%) compared with the meal plan groups (13%, p = 0.003).

Barriers to weight management. The lack of affordable, accessible transportation represents a significant barrier for both attending on-site meetings required in traditional weight management programs, and for engaging in PA (30, 60-62). Dr. Nary and colleagues completed a web-based needs assessment survey of 182 practitioners who provide services to adults with physical disabilities through Centers for Independent Living (63). Transportation was reported as the most frequent barrier to health care by 89% of respondents, while 78% and 65% reported their consumers could use information on diet and nutrition, and weight monitoring, respectively. Adults with MRDs may have a limited understanding as to what constitutes a healthy diet, and experience difficulty with food shopping and meal preparation (64-66). A survey of 1,096 women with disabilities indicated that ~33% experienced barriers to achieving optimal nutrition. Being too tired to cook was most frequently reported (~55%) (67). In addition to barriers to PA experienced by the general population, e.g., lack of time and motivation, adults with MRDs are confronted with inaccessible recreational facilities, lack of affordable and accessible fitness equipment, and poor infrastructure (lack of sidewalks and curb cuts, narrow/damaged sidewalks etc.) (62, 68-70). As described in detail in subsequent sections, remote or home visit delivery, and the use of a diet, that simplifies food shopping and preparation, will eliminate/reduce these barriers in the proposed interventions.

### **RATIONALE**

Premise/summary of significance/impact. The premise of this study is that adults with MRDs represent a sizeable and growing segment of the population, with a high prevalence of overweight/obesity, and limited empirically based options for effective weight management. The majority of weight loss trials (60%) that have included both ambulatory and non-ambulatory adults with MRDs have used 1-group, pre-post designs, in small samples ( $n \le 16$ ), over relatively short time frames (≤ 20 wks.) (55-57). These trials have shown unimpressive results in terms of both mean weight loss, and the percentage of participants losing ≥ 5% of baseline weight. In contrast to previous work, results from our 12 mo. trial in adults with MRDs suggested the potential effectiveness of a simplified dietary approach (eSLD) combined with monthly, home visit behavioral sessions (58). Although these results are encouraging, alternative strategies to provide weight management to greater numbers of adults with MRDs, potentially improve outcomes, and reduce costs are warranted. The proposed two-arm randomized trial will compare weight loss (6 mos.) and maintenance (12 mos.) between an individual home visit intervention (IH), using a protocol similar to our previous trial, and an intervention delivered remotely via video conferencing to groups of overweight/obese adults with MRDs in their homes (GR), and utilizing available technology for self-monitoring and increasing PA. We expect clinically meaningful weight loss in both intervention arms, i.e. ≥ 5%, with significantly greater weight loss in the GR arm. If successful, the GR intervention has the potential to be implemented in a variety of settings to provide effective weight management for adults with MRDs at a reasonable cost.

## STUDY TYPE AND DESIGN

We propose a 2-arm randomized trial (group remote (GR) vs. individual home visit (IH)) using intent-to-treat principles, to compare body weight following weight loss (6 mos.) and maintenance (18 mos.) in overweight/obese adults with MRDs. interventions will be delivered by trained health educators and will include behavioral sessions, a reduced energy diet (eSLD), increased PA, and self-monitoring of weight using electronic scales. The GR arm will be delivered via video conferencing (Zoom™ software) on a tablet computer (iPad mini) with selfmonitoring of diet and PA using commercially available technologies. Participants in the IH arm will self-monitor diet and PA using paper and pencil records. Due to COVID-19, all Cohort 1 IH intervention meetings will be held by phone per CDC social distancing recommendations. Participants are asked to send pictures of the tracking sheets to the health educator prior to the phone meeting. The primary outcome (weight) will be assessed during home visits at baseline (mo. 0), following weight loss (6 mos.), during (12 mos.) and at the end of maintenance (18 mos.). Our group has experience with all proposed intervention components and outcome assessments from previously completed (44, 58, 71, 78, 88, 89) or on-going trials (DK83589, HD79642). The following design attributes, described in detail subsequently, ensure the scientific rigor of the proposed trial: 1) Randomized design with equal allocation to groups, with allocation assignment concealed. 2) Adequate statistical power to address the primary aim. 3) Strategies to ensure the recruitment of sufficient participants to achieve our desired sample size. 4) Retention/incentive strategies to reduce loss to follow-up. 5) Controlling for attention by maintaining equal contact in both groups. 6) Secondary/exploratory aims to maximize the use of data, e.g., analysis to examine the impact of process variables/participant characteristics on

weight change. 7) The use of a theory-based intervention delivered by trained health educators. 8) Delivery of both intervention arms by the same health educator to cohorts of participants to minimize potential health educator effects. 9) Procedures to ensure intervention fidelity. 10) Assessments completed by trained staff blind to intervention arm. 11) Evaluation of staff interrater reliability for all physical assessments (2-3 times/yr.). 12) A novel assessment of diet to improve data quality. 13) Structured interviews at both 6 and 18 mos. to gather information that might be useful in improving the intervention and/or implementing the intervention in settings serving individuals with MRDs.

### SUBJECT CRITERIA

Primary care physician (PCP) clearance will be required of all participants. To enhance generalizability, individuals receiving treatment for prevalent chronic diseases, or with risk factors such as hypertension, tobacco use, lipid abnormalities, DM2, etc., will be allowed to participate with PCP clearance.

Inclusion criteria: 1) A permanent MRD (≥ 1 yr. duration) requiring the use of a wheelchair or resulting in the inability to walk 0.25 miles without stopping, with or without assistive devices, as documented by 7 items from the NHANES Physical Function Survey (113), and confirmed by the PCP. Individuals with MRDs, associated with, but not limited to spinal cord injury (SCI), spina bifida, multiple sclerosis, cerebral palsy, stroke, muscular dystrophy, and lower limb amputation will be included. 2) Age 18 and older. Weight management for younger individuals requires different behavioral strategies. 3) Body mass index (BMI) >25 kg/m² and body weight ≤400lbs. Individuals with a BMI <25 kg/m² are not overweight, and individuals over 400lbs may require more aggressive weight loss interventions, e.g., surgery, medication, etc. We are aware of the difficulty in the assessment of BMI, and issues related to the use of BMI for classifying overweight/obesity in individuals with SCI or amputations (114-116). Thus, in questionable cases we will defer to the PCP regarding eligibility based on weight status. 4) Wireless internet access in the home.

Exclusion criteria: 1) Unable to participate in light-to-moderate intensity PA, e.g., seated aerobics, resistance exercise, or physically unable to use the iPad. 2) Participation in a structured weight loss or exercise program in the previous 6 mos. These proximal experiences may influence this trial. 3) Current exercise (> 3, 30-min bouts of planned exercise/wk.) 4) Not weight stable (±4.6 kg) for 3 mos. prior to intake. 5) Unwilling to be randomized. 6) Pregnancy during the previous 6 mos., currently lactating, or planned pregnancy in the following 18 mos. 7) Serious medical risk, e.g., cancer, recent heart attack, stroke as determined by the PCP. 8) Current use of antipsychotics, untreated depression, or other psychiatric illness that would preclude participation in weight management, as determined by the PCP. Psychiatric comorbidity may limit the benefits from health education. Addressing psychiatric issues is beyond the scope of this study. 9) Cognitive, visual, or hearing impairments that may interfere with compliance to the study protocol as determined by the PCP. 10) Adherence to specialized diets, e.g., food allergies, vegetarian, macrobiotic. 11) Binge (Binge Eating Scale) (117) or other eating disorders (EATs-26) (118). 12) Living in the same household as another study participant.

### INTERVENTION DESCRIPTION

Orientation. Health educators will conduct home visits (~90 min) with all participants prior to initiating the intervention to provide a detailed description of both the dietary (eSLD) and PA components of the intervention and delivery formats (remote or home visit). All participants will be provided with an iPad mini tablet computer and electronic wireless scales. Access to nonstudy related materials, e.g., web browsing, app store etc., will be blocked on all iPads until completion of the study. iPads for the GR arm will be pre-loaded with the video conferencing (Zoom<sup>TM</sup> software), the Lose It! and Fitbit applications, and behavioral session materials (described later). Participants in the IH arm will be provided with hard copies of the intervention materials and will be shown how to self-monitor diet and PA using hard copy records. During orientation, both intervention arms will receive a tutorial on the use of the iPad and electronic scales, and procedures for making digital photographs of meals, to be used in the assessment of dietary intake (described in assessment section). Participants in the GR arm will be oriented to the video conferencing software and both the Lose it! and Fitbit apps/devices used for selfmonitoring diet and PA. Time will be allotted for practice and questions. Per inclusion/exclusion criteria, those unable to perform these tasks will be ineligible. Tutorials describing trouble shooting for common technical problems, e.g., internet connectivity, data entry using Fitbit, Lose It!, will be loaded on the iPad. Technical issues can also be resolved during behavioral sessions, or by contacting research staff by phone or email. The GR arm will be provided with an HDMI adaptor allowing video conference sessions to be displayed on a larger TV screen, if desired. Reminders regarding upcoming behavioral/PA sessions etc., or to prompt participants in the GR arm who are non-compliant with the study protocol, will be sent via the iPad.

<u>Diet (0-6 mos.)</u>. The original SLD, developed for use in children (59), categorizes foods by energy content. The SLD is easy to understand and implement when compared with a meal plan diet. Meal plan diets require choosing appropriate foods from an unlimited array of options, making it difficult to prepare a nutritionally adequate reduced energy diet on a consistent basis. We will "enhance" the Stop Light Diet (eSLD) using a combination of commercially available portion-controlled meals (PCMs- meals/shakes) and fruits and vegetables. PCMs include nutritional information on the label (calories, fat, protein etc.) making it easier to adhere to specific energy and nutrient prescriptions. Participants will be asked to consume a minimum daily total of 2 meals (~200 to 300 kcal each, saturated fat ≤ 3g), 3 shakes (~100 kcal each), five 1-cup servings of fruits/vegetables, and ad libitum non-caloric beverages. Participants will be asked to purchase PCMs (meals/shakes) from a list meeting these caloric/fat requirements, as well as fruits/vegetables, and non-caloric beverages. The recommended PCMs are affordable and available at most grocery stores at a cost of \$2-\$4 each, which may be an important consideration for individuals with MRDs where household income is often low (1). Dr. Ptomey, RDN will assure all diets are energy and nutritionally adequate, and will follow the AND Evidence Library Nutritional Guidelines for individuals with SCI (121).

<u>Diet (7-18 mos.).</u> During weight maintenance participants will be encouraged to continue using the eSLD, or transition to a meal plan, or combination eSLD/meal plan diet. At the end of the weight loss phase (mo. 6) counseling will include tips for complying with a conventional diet, i.e., meal planning, food shopping, meal preparation, portion control, etc.

Energy intake-weight loss (0-6 mos.). Energy intake will be prescribed at 1,200-1,500 kcal/d for women and 1,500-1,800 kcal/d for men as recommended by current weight management quidelines from the American Heart Association/American College of Cardiology/The Obesity Society (53). We are aware that these recommendations were not designed specifically for adults with MRDs, and may be inappropriate for individuals with SCI due to variable reductions in energy expenditure associated with level and duration of injury, adrenergic function, and fatfree-mass (123-126). We will estimate energy needs for individuals with paraplegia (27.9 kcal/kg/d) and tetraplegia (22.7 kcal/kg/d) as recommended by Cox et al (127) with upward adjustment for individuals with pressure ulcers as suggested by the AND Evidence Library Nutritional Guidelines for individuals with SCI (121). The proposed levels of energy intake provide a reasonable starting point, and will be adjusted based on the observed weight change and participant feedback regarding hunger/satiation. Participants for whom additional weight loss would be contraindicated, e.g., BMI of ≤ 22 kg/m<sup>2</sup> or losing > 20% of baseline weight, will be placed on a weight maintenance diet at any time during the intervention. Those who continue to lose weight will be referred to appropriate health professionals/agencies, and may be dismissed from the trial if necessary.

Energy intake-weight maintenance (7-18 mos.). Energy intake for weight maintenance will be based on the RMR equation of Mifflin-St Jeor (128) adjusted for activities of daily living (RMR x 1.4-1.6) as participants will have a routine PA program. As described for weight loss, we will use the energy need estimates of Cox et al (127) and the AND Evidence Library for individuals with SCI (121). In our experience, some participants not meeting their weight loss goals (0-6 mos.) will volitionally attempt additional weight loss during maintenance (7-18 mos.); which will not be encouraged or discouraged. Participants experiencing weight gain will be counseled to improve compliance with the diet and PA protocols. We have successfully employed this approach for prescribing energy intake for weight loss/maintenance in previous trials in adults with MRDs (58), and in adults with (73, 89), and without IDD (71).

Behavioral session/frequency/duration (Table 1). GR arm. Behavioral sessions (10-15 individuals) will be conducted using video conferencing (Zoom<sup>TM</sup> software) 2/mo. during weight loss and the first 6 mos. of maintenance (mos. 0-12), and 1/mo. during the last 6 mos. of maintenance (mos. 13-18). IH arm. Behavioral sessions will be conducted with individual participants during home visits. Behavioral sessions in the IH arm will follow the same frequency as the GR arm and will occur 2/mo. during weight loss and the first 6 mos. of maintenance (mos. 0-12), and 1/mo. during the last 6 mos. of maintenance (mos. 13-18). Meeting duration will be 45-60 min. for both groups across the intervention. Due to COVID-19, all Cohort 1 IH intervention meetings will be held by phone per CDC social distancing recommendations. Participants are asked to send pictures of the tracking sheets to the health educator prior to the phone meeting

<u>Behavioral session content-weight loss.</u> Behavioral sessions will be identical between groups and will include a review of participants self-monitored data for diet, PA, and weight recorded since the previous session, a question to generate discussion regarding diet and PA, a lesson on a weight management topic, and an experiential learning assignment requiring problem solving or the practice of behavioral strategies, to be completed prior to the next session. Lessons will also include topics such as cost and time efficient strategies for food shopping and

preparation, specific strategies for increasing daily PA and decreasing sedentary time, and maintaining adequate hydration, eating away from home etc., with examples and discussion questions specific to individuals with MRDs.

<u>Behavioral session content-weight maintenance.</u> Behavioral sessions during maintenance will focus on planning and following a meal plan diet, with or without incorporation of PCMs, and cardinal behaviors for successful weight maintenance, such as self-monitoring, regular PA, eating on weekends/vacations, and controlling energy intake on special occasions and holidays, etc.

PA prescription. We will target 150 min./wk. of moderate-intensity aerobic activity (3-6 METs), and 2 d/wk. of resistance training (RT) for intervention arms as recommended for adults with/without disabilities by the American College of Sports Medicine (129) and the U.S. Department of Health and Human Services (130). This level of exercise is well within the capability of adults with MRDs, including those with SCI (131, 132); however, participants unable to complete 150 min. /wk. will be encouraged to exercise to their individual capacities. We recognize that 150 min./wk. is less than the 300 min./wk. recommended for weight management (133). However, given the limits to the levels of energy expenditure, from what will be predominantly upper extremity exercise, and the increased potential for overuse injuries with higher volumes of exercise (134), we felt that 300 min./wk. would be unrealistic in this sample. Aerobic exercise will progress from 60 min/wk. (3 d/wk., 20 min./d) to 150 min. /wk. (5 d/wk., 30 min./d) at the beginning of mo. 4, and remain at 150 min./wk. through mo. 18. RT (3 sets/8-10 reps, 4-5 exercises) using resistance bands (8 levels) provided by the study (Theraband, Akron OH) will be prescribed. RT, as well as a stretching regime, will focus on scapular stabilizers and posterior shoulder muscles, and major lower extremity muscles for participants with this capability. During the first 2 wks., participants will use a band that provides a resistance allowing completion of 3 sets with minimal fatigue. Resistance will be increased to the next level at wk. 3, and increased subsequently, when participants are able to complete 3 sets of 8-10 reps with minimal fatigue. The negative health consequences of sedentary behavior (135, 136) may be especially relevant for individuals with MRDs (62, 137). Therefore, strategies for decreasing sedentary time, such as increasing sit-to-stand transitions and standing time, in those who are able, and increasing non-exercise upper extremity activity, e.g., daily light activities for wheelchair users, will be recommended.

<u>PA delivery.</u> Participants in the GR arm will be asked to attend 30-min group exercise sessions conducted using video conferencing (Zoom<sup>™</sup> software) 2 x/wk. during weight loss (0-6 mos.) and 1x/wk. during maintenance (7-18 mos.) Exercise sessions will be conducted in conjunction with behavioral sessions when schedules coincide. In such cases the total session time (behavioral+exercise) will not exceed 60 min. Group sessions will include a warm-up, 20 min. of moderate intensity aerobic activity, 10 min of RT, and stretching and cool-down. Exercise sessions will include individuals with a range of functional abilities, e.g., wheelchair users/ambulatory. Dr. Greene, an adapted PA specialist, will modify activities, as necessary, to insure they are applicable for all participants. Our trial in adolescents with IDD demonstrated the feasibility of the home-based group video conference approach for delivering exercise to groups varying widely in physical abilities (preliminary studies). Group sessions will provide 40 minutes of the 150 min./wk. recommendation for aerobic activity. To assist participants in both study

arms in meeting the 150 min./wk. goal, all group sessions will be video recorded and uploaded remotely to participant's iPads where they can be accessed for use at any time. In addition, information regarding exercise resources available from the National Center on Health, Physical Activity and Disability, Craig Hospital, and the Christopher and Dana Reeve Foundation will be pre-loaded on the iPad of participants in all study groups. *The IH arm* will be asked to complete the exercise recommendations on their own, as is customary in standard care weight management. Participants in the *IH* arm will receive brief (5-10 mins.) support/problem solving phone calls (1x.wk.) and iMessages (1x/wk) from the health educator an approach that has been shown to increase exercise in adults with MRDs (44).

#### **OUTCOME MEASURES**

<u>Weight/Height: Ambulatory participants.</u> Weight will be measured in duplicate with a portable, calibrated digital scale. (Model #PS6600, Befour, Saukville, WI.). Standing height will be measured in duplicate with a portable stadiometer (Model #IP0955, Invicta Plastics Limited, Leicester, UK).

<u>Weight/Height: Wheelchair users</u>. Weight will be measured in duplicate using a portable calibrated, digital wheelchair scale (Model MX420, Befour, Saukville, WI.). Participant weight will be calculated as participant + chair weight minus chair weight. Digital photos of the chair will be obtained at baseline to ensure that the same chair (and accessories) is used for subsequent assessments, thus negating the need for repeated assessments of chair weight. Supine height will be assessed with a metal tape with legs outstretched and feet in dorsiflexion. If contractures prevent assessment of supine height, we will estimate total height based on knee height as described by Froehlich-Grobe et al (87).

<u>Waist circumference</u> will be assessed using the procedures described by Lohman et al. (144). Three measurements will be obtained with the outcome recorded as the average of the closest 2 measures.

<u>Blood pressure</u> will be obtained with an automated sphygmomanometer (DinaMap ProCare 100, General Electric) using the NHANES blood pressure protocol (145).

<u>Quality of life</u> will be assessed with the SF-36E, a version of the SF-36 (147, 148) in which the PA section has been modified for individuals with MRDs (149). The SF-36E has acceptable psychometric properties (149).

<u>Demographics</u>. In addition to basic demographics/health history, we will assess type/duration of MRD, living arrangement (alone/with others), employment status, and level of responsibility for food shopping and preparation.

<u>Cost analysis (Dr. Lee)</u>. A cost analysis may be considered premature. However, this may be the only opportunity we will have to complete such analyses, which can be done at minimal expense, in a large sample of adults with MRDs. Based on a previous weight loss trial (71) we expect higher costs associated with health educator travel required in the *IH* arm. Mean weight loss at 6 mos. will serve as our measure of effectiveness. We expect greater weight loss and lower costs in the *GR* compared with the *IH* arms (150). We will then calculate the cost per additional kg of weight loss. Contingent valuation analysis, in which participants express preferences for programs, will be used to examine the perceived worth of the *GR* and *IH* formats at 6 and 18 mos.(151). Conditional logistic regressions, with adjustments for clustering by health educator, will be used to analyze how differences in client attributes, anticipated costs, and anticipated gains affect preferences for the 2 intervention arms. The cost perspective for all

analyses will be societal. We will collect data on both program and participant costs prospectively. The gold standard for measuring cost is a time study based on a validated flowchart (152, 153). We will validate flowcharts for both study arms and use time studies to estimate health educator time, and program records to measure cost of supplies. Participant time, valued at the local median hourly wage, is also a component of intervention costs (154) as time devoted to an intervention cannot be used for work or leisure. These costs may be half of the total costs (155, 156) and will be gathered via survey (157).

Energy Expenditure of Remote Exercise Sessions (optional). Energy expenditure of the remote sessions will be assessed in a volunteer sample using a previously validated portable, open-circuit indirect calorimeter (Cosmed, Italy) which measures breath-by-breath ventilation, expired oxygen, and carbon dioxide. The flow turbine will be calibrated using a 3.0-L syringe. The lightweight (~1.5 kg) portable system will be attached by a harness around the waist and shoulders of the participant before each assessment. During exercise sessions, participants will breathe into a facemask that directs air into the unit housing the O2 and CO2 analyzers. Data will be retrieved for analysis via a serial port interface and software provided with the calorimeter, and aggregated over 20-second epochs for the calculation of 1-min averages. MET levels will be age corrected using the Schofield equation (88) as recommended by McMurray et al (89). Participants will be asked to wear wrist ActiGraphs during the assessment for comparison of physical activity levels between devices.

## SAMPLE SIZE, STATISTICAL METHODS, AND POWER CALCULATION

**Power/sample size.** The mean 6 mo. weight loss in our completed trial in adults with MRDs, using a protocol similar to the *IH* arm in the proposed trial, i.e., eSLD and behavioral counseling delivered by monthly home visits, was 5.5 kg (58). This does not reach the 8.5 kg ( $\sim$ 5%) average 6 mo. weight loss defined as clinically meaningful by current weight management guidelines (53). We expect 6 mo. weight loss in the *GR* arm, which includes weekly group counseling and group exercise, will reach or exceed 8.5 kg. To detect a clinically meaningful difference of 3 kg (133, 176-180) in 6 mos. weight loss between the *IH* and *GR* arms, with 80% power and a type 1 error rate of 0.05, assuming a common standard deviation of 6 kg, will require 64 participants/group. Secondarily, we will have 70% power to detect a 3 kg difference in a completer analysis with an attrition rate of 20%; however, we expect attrition will be lower based on experience (71, 78, 181), and our use of retention/incentive strategies to minimize loss to follow-up. Thus, a sample of 64/group will provide adequate power for both our primary intent-to-treat analysis with imputed missing data (power = 80%) and our secondary completer only analysis (70%).

**Analysis plans.** <u>Primary aim</u> will use a 2-sample independent t-test to compare 6 mo. weight loss between the 2 intervention arms in both an intent-to-treat, and completer only analysis. Procedures for handling missing data are described below. We will examine the impact of baseline characteristics (age, sex, race/ethnicity, weight, type of MRD, wheelchair use, employment status, living situation, food shopping and preparation) on weight change using linear regression controlling for treatment. We will examine the main effects of each of these variables, as well as the potential interaction effect with treatment.

<u>Secondary aim 1, a comparison of 18 mo. weight loss,</u> will mirror the analysis for the primary aim. We will use a 2-sample t-test to compare weight change (0-18 mos.) between the 2 intervention arms. Mixed linear models will be used to compare weight change from 0-18 mos.

between intervention arms controlling for intervention arm and baseline weight. We anticipate greater loss to follow-up over time; however, we expect data to be missing at random. Under this assumption, mixed linear models will provide unbiased treatment comparisons. We will assume an autoregressive correlation structure of the dependent variable (weight) over time, and evaluate the potential for time-by-treatment interactions.

<u>Secondary aim 2, a between arm comparison of the proportion of participants achieving  $\geq 5\%$  weight loss (0-18 mos.)</u> will be evaluated using a chi-square test. Participants without an 18 mo. weight will be classified as not meeting the  $\geq 5\%$  weight loss goal. We will also examine the impact of baseline characteristics, as previously defined, on 18 mo. weight loss using logistic regression.

<u>Secondary aims 3 and 4, between arm comparison of change in risk factors and quality of life</u> (0-6 and 0-18 mos.) will be evaluated using a 2-sample t-test.

Exploratory <u>aims</u> will examine the influence of the following on weight loss at 6 mos.: behavioral session attendance, compliance with the recommendations for diet (energy intake, number of meals/shakes, servings of fruits/vegetables), PA (min of moderate-vigorous PA, min sedentary time), self-monitoring of diet and PA, sleep, and medications assessed over the time period of interest, i.e. (0-6 and 0-18 mos.) and the change in self-efficacy for PA and dietary change, dietary self-regulation, social support for diet/PA, and barriers to PA from 0-6 mos. We will examine the influence of these factors as covariates, in addition to treatment, on weight loss at 6 mos. As we have 128 observations with a rule of thumb of at least 30 observations for each variable in the model, judicious model selection will be completed as we can only expect to identify ~4 variables that are related to weight loss in a single model. First, we will assess if these variables differ by treatment at the 0.10 level and if they do they will be considered for future modeling. If in a two-factor model, the variable and treatment have a potential interaction at the 0.10 level that interaction will be considered for future modeling. Subsequently, the main effects and interaction effects along with treatment will be examined in a joint model. Given the pitfalls of forward and backward selection, we will utilize best subsets criteria based upon Mallow's Cp statistic to produce the most parsimonious and least biased model of weight loss at 6 months. This should allow us to identify what variables most highly influence our outcome along with treatment and/or the mechanism(s) of action that are impacting weight loss. We will do the same for weight loss at 18 months, as this measure may have similar or different variables that impact this long-term outcome.

**Missing Data/ imputation.** All analyses will be based on intent-to-treat principles and missing data for analyses of the primary aim will be imputed; therefore, oversampling for attrition is not needed. We will determine if the proportion of participants lost to follow-up differs by treatment. If so, we will determine if there are differences in demographic characteristics (sex, age, baseline weight, p < 0.05) between completers and those lost to follow-up. If missing data are related to treatment and/or these demographic characteristics, we will use model based multiple imputation; otherwise, we will use traditional multiple imputation. Statistical analysis will be completed with SAS version 9.4 or higher.

### REFERENCES

- 1. Courtney-Long EA, Carroll DD, Zhang Q, C., Stevens AC, Griffin-Blake S, Armour BS, Campbell VA. Prevalence of disability and disability type amound adults United States, 2013. MMWR. 2015;64(29):777-83.
- 2. Brault MW. Americans with Disabilities: 2010 Current Population Reports. Washington, DC: US Census Bureau; 2012. p. 40-131.
- 3. Stevens AC, Carroll DD, Courtney-Long EA, Zhang QC, Sloan ML, Griffin-Blake S, Peacock G. Adults with One or More Functional Disabilities United States, 2011-2014. MMWR Morbidity and mortality weekly report. 2016;65(38):1021-5. Epub 2016/09/30. doi: 10.15585/mmwr.mm6538a1. PubMed PMID: 27684532.
- 4. Liou TH, Pi-Sunyer FX, Laferrere B. Physical disability and obesity. Nutrition reviews. 2005;63(10):321-31. Epub 2005/11/22. PubMed PMID: 16295145.
- 5. lezzoni LI, Kurtz SG, Rao SR. Trends in U.S. adult chronic disability rates over time. Disability and health journal. 2014;7(4):402-12. Epub 2014/09/17. doi: 10.1016/j.dhjo.2014.05.007. PubMed PMID: 25224980; PMCID: Pmc4167341.
- 6. Lauer EA, Houtenville AJ. Annual Disability Statistics Compendium: 2016. Durham, NH: University of New Hampshire, Institute on Disability, 2017.
- 7. Brucker DL, Houtenville AJ. People with disabilities in the United States. Archives of physical medicine and rehabilitation. 2015;96(5):771-4. Epub 2015/03/12. doi: 10.1016/j.apmr.2015.02.024. PubMed PMID: 25757791.
- 8. Carroll DD, Courtney-Long EA, Stevens AC, Sloan ML, Lullo CV, S.N., Fox MH, Armour BS, Campbell VA, Brown DR, Dorn JM. Vital Signs: Disability and physical activity United States, 2009-2012. MMWR. 2014;63(18):407-13.
- 9. Burki TK. More hurdles: exercise for people with disabilities. The Lancet Diabetes & Endocrinology. 2015;3(1):14. Epub 2014/12/10. doi: 10.1016/s2213-8587(14)70245-1. PubMed PMID: 25488099.
- 10. Havercamp SM, Scott HM. National health surveillance of adults with disabilities, adults with intellectual and developmental disabilities, and adults with no disabilities. Disability and health journal. 2015;8(2):165-72. Epub 2015/01/18. doi: 10.1016/j.dhjo.2014.11.002. PubMed PMID: 25595297.
- 11. Ginis KA, Latimer AE, Arbour-Nicitopoulos KP, Buchholz AC, Bray SR, Craven BC, Hayes KC, Hicks AL, McColl MA, Potter PJ, Smith K, Wolfe DL. Leisure time physical activity in a population-based sample of people with spinal cord injury part I: demographic and injury-related correlates. Archives of physical medicine and rehabilitation. 2010;91(5):722-8. Epub 2010/05/04. doi: 10.1016/j.apmr.2009.12.027. PubMed PMID: 20434609.
- 12. Littman AJ, Boyko EJ, Thompson ML, Haselkorn JK, Sangeorzan BJ, Arterburn DE. Physical activity barriers and enablers in older Veterans with lower-limb amputation. Journal of rehabilitation research and development. 2014;51(6):895-906. Epub 2014/10/31. doi: 10.1682/jrrd.2013.06.0152. PubMed PMID: 25356624.
- 13. Usuba K, Oddson B, Gauthier A, Young NL. Leisure-Time Physical Activity in adults with Cerebral Palsy. Disability and health journal. 2015;8(4):611-8. Epub 2015/07/05. doi: 10.1016/j.dhjo.2015.05.006. PubMed PMID: 26141088.
- 14. Xu B, Houston D, Locher JL, Zizza C. The association between Healthy Eating Index-2005 scores and disability among older Americans. Age and ageing. 2012;41(3):365-71. Epub 2011/12/16. doi: 10.1093/ageing/afr158. PubMed PMID: 22169770.
- 15. An R, Chiu CY, Zhang Z, Burd NA. Nutrient intake among US adults with disabilities. Journal of human nutrition and dietetics: the official journal of the British Dietetic Association. 2015;28(5):465-75. Epub 2014/09/23. doi: 10.1111/jhn.12274. PubMed PMID: 25233949.

- 16. Froehlich-Grobe K, Lee J, Washburn RA. Disparities in obesity and related conditions among Americans with disabilities. American journal of preventive medicine. 2013;45(1):83-90. Epub 2013/06/26. doi: 10.1016/j.amepre.2013.02.021. PubMed PMID: 23790992.
- 17. Chevarley FM, Thierry JM, Gill CJ, Ryerson AB, Nosek MA. Health, preventive health care, and health care access among women with disabilities in the 1994-1995 National Health Interview Survey, Supplement on Disability. Women's health issues: official publication of the Jacobs Institute of Women's Health. 2006;16(6):297-312. Epub 2006/12/26. doi: 10.1016/j.whi.2006.10.002. PubMed PMID: 17188213.
- 18. Coyle CP, Santiago MC, Shank JW, Ma GX, Boyd R. Secondary conditions and women with physical disabilities: a descriptive study. Archives of physical medicine and rehabilitation. 2000;81(10):1380-7. Epub 2000/10/13. doi: 10.1053/apmr.2000.9169. PubMed PMID: 11030504.
- 19. Dixon-Ibarra A, Horner-Johnson W. Disability status as an antecedent to chronic conditions: National Health Interview Survey, 2006-2012. Preventing chronic disease. 2014;11:130251. Epub 2014/02/01. doi: 10.5888/pcd11.130251. PubMed PMID: 24480632; PMCID: Pmc3917726.
- 20. Reichard A, Stolzle H, Fox MH. Health disparities among adults with physical disabilities or cognitive limitations compared to individuals with no disabilities in the United States. Disability and health journal. 2011;4(2):59-67. Epub 2011/03/23. doi: 10.1016/j.dhjo.2010.05.003. PubMed PMID: 21419369.
- 21. Hollar DW, Jr., Lewis JS. Heart age differentials and general cardiovascular risk profiles for persons with varying disabilities: NHANES 2001-2010. Disability and health journal. 2015;8(1):51-60. Epub 2014/09/10. doi: 10.1016/j.dhjo.2014.07.007. PubMed PMID: 25200711.
- 22. Hollar D. Cross-sectional changes in patterns of allostatic load among persons with varying disabilities, NHANES: 2001-2010. Disability and health journal. 2013;6(3):177-87. Epub 2013/06/19. doi: 10.1016/j.dhjo.2013.01.009. PubMed PMID: 23769476.
- 23. Washburn RA, Figoni SF. High density lipoprotein cholesterol in individuals with spinal cord injury: the potential role of physical activity. Spinal cord. 1999;37(10):685-95. Epub 1999/11/11. PubMed PMID: 10557124.
- 24. Stevens A, Courtney-Long E, Gillespie C, Armour BS. Hypertension among US adults by disability status and type, National Health and Nutrition Examination Survey, 2001-2010. Preventing chronic disease. 2014;11:E139. Epub 2014/08/15. doi: 10.5888/pcd11.140162. PubMed PMID: 25121351; PMCID: Pmc4133509.
- 25. Forman-Hoffman VL, Ault KL, Anderson WL, Weiner JM, Stevens A, Campbell VA, Armour BS. Disability status, mortality, and leading causes of death in the United States community population. Medical care. 2015;53(4):346-54. Epub 2015/02/27. doi: 10.1097/mlr.000000000000321. PubMed PMID: 25719432.
- 26. Majer IM, Nusselder WJ, Mackenbach JP, Klijs B, van Baal PH. Mortality risk associated with disability: a population-based record linkage study. American journal of public health. 2011;101(12):e9-15. Epub 2011/10/25. doi: 10.2105/ajph.2011.300361. PubMed PMID: 22021307; PMCID: Pmc3222426.
- 27. Shields M, Gorber SC, Tremblay MS. Effects of measurement on obesity and morbidity. Statistics Canada-Health Reports. 2008;19(2):1-8.
- 28. Hattori A, Sturm R. The obesity epidemic and changes in self-report biases in BMI. Obesity (Silver Spring, Md). 2013;21(4):856-60. Epub 2013/05/29. doi: 10.1002/oby.20313. PubMed PMID: 23712990.

- 29. Froehlich-Grobe K, Nary DE, VanSciver A, Washburn RA, Aaronson L. Truth be told: evidence of wheelchair users' accuracy in reporting their height and weight. Archives of physical medicine and rehabilitation. 2012;93(11):2055-61. Epub 2012/05/23. doi: 10.1016/j.apmr.2012.05.005. PubMed PMID: 22609118; PMCID: Pmc3562126.
- 30. Locatelli SM, Gerber BS, Goldstein B, Weaver FM, LaVela SL. Health care provider practices, barriers, and facilitators for weight management for individuals with spinal cord injuries and disorders. Topics in spinal cord injury rehabilitation. 2014;20(4):329-37. Epub 2014/12/06. doi: 10.1310/sci2004-329. PubMed PMID: 25477746; PMCID: Pmc4252133.
- 31. Liusuwan RA, Widman LM, Abresch RT, Johnson AJ, McDonald CM. Behavioral intervention, exercise, and nutrition education to improve health and fitness (BENEfit) in adolescents with mobility impairment due to spinal cord dysfunction. The journal of spinal cord medicine. 2007;30 Suppl 1:S119-26. Epub 2007/09/19. PubMed PMID: 17874697; PMCID: Pmc2031996.
- 32. Fitzgerald SJ, Kelleher AR. Mobility challenges in individuals with a spinal cord injury with increased body weight. Topics in Spinal Cord Injury Relabilitation. 2007;12(4):54-63.
- 33. Gater DR, Jr. Obesity after spinal cord injury. Physical medicine and rehabilitation clinics of North America. 2007;18(2):333-51, vii. Epub 2007/06/05. doi: 10.1016/j.pmr.2007.03.004. PubMed PMID: 17543776.
- 34. Holmgren M, Lindgren A, de Munter J, Rasmussen F, Ahlstrom G. Impacts of mobility disability and high and increasing body mass index on health-related quality of life and participation in society: a population-based cohort study from Sweden. BMC public health. 2014;14:381. Epub 2014/04/20. doi: 10.1186/1471-2458-14-381. PubMed PMID: 24742257; PMCID: Pmc4036728.
- 35. Karpur A, Bruyere SM. Health care expendiure among people with disabilities: Potential role of workplace health promoion and implications for rehabilitation counseling. Rehabilitation Counseling Bulletin. 2012;56(1):7-22.
- 36. Anderson WL, Wiener JM, Khatutsky G, Armour BS. Obesity and people with disabilities: the implications for health care expenditures. Obesity (Silver Spring, Md). 2013;21(12):E798-804. Epub 2013/06/28. doi: 10.1002/oby.20531. PubMed PMID: 23804319; PMCID: PMC4494729.
- 37. The Future of Disability in America. Washington, DC: Institute of Medicine, Committee on Disability in America, 2007.
- 38. The Current State of Health Care for People with Disabilities. Washington, DC: National Council on Disability, 2009.
- 39. United States Department of Health and Human Services, Healthy People 2010, 2nd ed. Washington, DC. 2000.
- 40. Healthy People 2020. Washington, DC: U.S. Department of Health and Human Services, Office of Disease Prevention and Health Promotion. p.
- https://www.healthypeople.gov/2020/topics-objectives/topic/disability-and-health Accessed 12/10/15.
- 41. Patient Protection and Affordable Care Act of 2010, PL 111-148. 2010. p. <a href="http://democrats.senate.gov/reform/patient-protection-affordable-care-act-as-passed.pdf">http://democrats.senate.gov/reform/patient-protection-affordable-care-act-as-passed.pdf</a>. Accessed 11/7/2015.
- 42. Arbour-Nicitopoulos KP, Ginis KA, Latimer AE. Planning, leisure-time physical activity, and coping self-efficacy in persons with spinal cord injury: a randomized controlled trial. Archives of physical medicine and rehabilitation. 2009;90(12):2003-11. Epub 2009/12/09. doi: 10.1016/j.apmr.2009.06.019. PubMed PMID: 19969161.

- 43. Arbour-Nicitopoulos KP, Tomasone JR, Latimer-Cheung AE, Martin Ginis KA. Get in motion: an evaluation of the reach and effectiveness of a physical activity telephone counseling service for Canadians living with spinal cord injury. PM & R: the journal of injury, function, and rehabilitation. 2014;6(12):1088-96. Epub 2014/07/06. doi: 10.1016/j.pmrj.2014.05.018. PubMed PMID: 24990447.
- 44. Froehlich-Grobe K, Lee J, Aaronson L, Nary DE, Washburn RA, Little TD. Exercise for everyone: a randomized controlled trial of project workout on wheels in promoting exercise among wheelchair users. Archives of physical medicine and rehabilitation. 2014;95(1):20-8. Epub 2013/07/23. doi: 10.1016/j.apmr.2013.07.006. PubMed PMID: 23872080; PMCID: Pmc4610124.
- 45. Ravesloot C, Seekins T, Traci M, Boehm T, White G, Witten MH, Mayer M, Monson J. Living Well with a Disability, a Self-Management Program. MMWR supplements. 2016;65(1):61-7. Epub 2016/02/27. doi: 10.15585/mmwr.su6501a10. PubMed PMID: 26916136.
- 46. Ravesloot CH, Seekins T, Cahill T, Lindgren S, Nary DE, White G. Health promotion for people with disabilities: development and evaluation of the Living Well with a Disability program. Health education research. 2007;22(4):522-31. Epub 2006/10/13. doi: 10.1093/her/cyl114. PubMed PMID: 17032708.
- 47. Horner-Johnson W, Drum CE, Abdullah N. A randomized trial of a health promotion intervention for adults with disabilities. Disability and health journal. 2011;4(4):254-61. Epub 2011/10/22. doi: 10.1016/j.dhjo.2011.06.003. PubMed PMID: 22014673.
- 48. Abdullah N, Horner-Johnson W, C. D, Krahn GL, Staples E, Weisser J, Hammond L. Healthy Lifestyles for People with Disabilities. California Journal of Health Promotion. 2004;2(Special Issue):52-4.
- 49. Block P, Vanner EA, Keys CB, Rimmer JH, Skeels SE. Project Shake-It-Up: using health promotion, capacity building and a disability studies framework to increase self efficacy. Disability and rehabilitation. 2010;32(9):741-54. Epub 2010/03/23. doi: 10.3109/09638280903295466. PubMed PMID: 20302442.
- 50. Stuifbergen AK, Becker H, Blozis S, Timmerman G, Kullberg V. A randomized clinical trial of a wellness intervention for women with multiple sclerosis. Archives of physical medicine and rehabilitation. 2003;84(4):467-76. Epub 2003/04/12. doi: 10.1053/apmr.2003.50028. PubMed PMID: 12690582.
- 51. Ipsen C, Seekins T, Ravesloot C. Building the case for delivering health promotion services within the vocational rehabilitation system. Rehabilitation Counseling Bulletin. 2010;53:67-77.
- 52. Plow MA, Moore S, Husni ME, Kirwan JP. A systematic review of behavioural techniques used in nutrition and weight loss interventions among adults with mobility-impairing neurological and musculoskeletal conditions. Obesity reviews: an official journal of the International Association for the Study of Obesity. 2014;15(12):945-56. Epub 2014/10/01. doi: 10.1111/obr.12223. PubMed PMID: 25266576.
- 53. Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Journal of the American College of Cardiology. 2014;63(25 Pt B):2985-3023. Epub 2013/11/19. doi: 10.1016/j.jacc.2013.11.004. PubMed PMID: 24239920.

- 54. Rimmer JH, Wang E, Pellegrini CA, Lullo C, Gerber BS. Telehealth weight management intervention for adults with physical disabilities: a randomized controlled trial. American journal of physical medicine & rehabilitation / Association of Academic Physiatrists. 2013;92(12):1084-94. Epub 2013/11/22. doi: 10.1097/PHM.0b013e31829e780e. PubMed PMID: 24257266.
- 55. Chen Y, Henson S, Jackson AB, Richards JS. Obesity intervention in persons with spinal cord injury. Spinal cord. 2006;44(2):82-91. Epub 2005/08/17. doi: 10.1038/sj.sc.3101818. PubMed PMID: 16103891.
- 56. Betts AC, Froehlich-Grobe K. Accessible weight loss: Adapting a lifestyle intervention for adults with impaired mobility. Disability and health journal. 2017;10(1):139-44. Epub 2016/07/20. doi: 10.1016/j.dhjo.2016.06.004. PubMed PMID: 27431768.
- 57. Radomski MV, Finkelstein M, Hagel S, Masemer S, Theis J, Thompson M. A pilot wellness and weight managment program for individuals with spinal cord injury: Participants' goals and outcomes. Topics in spinal cord injury rehabilitation. 2011;17(2):59-69.
- 58. Reichard A, Saunders MD, Saunders RR, Donnelly JE, Lauer E, Sullivan DK, Ptomey L. A comparison of two weight management programs for adults with mobility impairments. Disability and health journal. 2015;8(1):61-9. Epub 2014/09/23. doi: 10.1016/j.dhjo.2014.08.002. PubMed PMID: 25242059.
- 59. Epstein L, Squires S. The Stoplight Diet for Children: An Eight-Week Program for Parents and Children. Boston, MA: Little Brown & Company; 1988.
- 60. Cardenas DD, Yilmaz B. Recruitment of spinal cord injury patients to clinical trials: Challenges and solutions. Topics in spinal cord injury rehabilitation. 2006;11(2):12-23.
- 61. Nosek MA, Hughes RB, Robinson-Whelen S, Taylor HB, Howland CA. Physical activity and nutritional behaviors of women with physical disabilities: physical, psychological, social, and environmental influences. Women's health issues: official publication of the Jacobs Institute of Women's Health. 2006;16(6):323-33. Epub 2006/12/26. doi: 10.1016/j.whi.2006.08.002. PubMed PMID: 17188215.
- 62. Rimmer JH, Schiller W, Chen MD. Effects of disability-associated low energy expenditure deconditioning syndrome. Exercise and sport sciences reviews. 2012;40(1):22-9. Epub 2011/10/22. doi: 10.1097/JES.0b013e31823b8b82. PubMed PMID: 22016146.
- 63. Living RaTCoC. Needs Assessment Report Lawrence, KS: 2015.
- 64. Bertoli S, Battezzati A, Merati G, Margonato V, Maggioni M, Testolin G, Veicsteinas A. Nutritional status and dietary patterns in disabled people. Nutrition, metabolism, and cardiovascular diseases: NMCD. 2006;16(2):100-12. Epub 2006/02/21. doi: 10.1016/j.numecd.2005.05.007. PubMed PMID: 16487910.
- 65. Tomey KM, Chen DM, Wang X, Braunschweig CL. Dietary intake and nutritional status of urban community-dwelling men with paraplegia. Archives of physical medicine and rehabilitation. 2005;86(4):664-71. Epub 2005/04/14. doi: 10.1016/j.apmr.2004.10.023. PubMed PMID: 15827915.
- 66. Mojtahedi MC, Boblick P, Rimmer JH, Rowland JL, Jones RA, Braunschweig CL. Environmental barriers to and availability of healthy foods for people with mobility disabilities living in urban and suburban neighborhoods. Archives of physical medicine and rehabilitation. 2008;89(11):2174-9. Epub 2008/11/11. doi: 10.1016/j.apmr.2008.05.011. PubMed PMID: 18996247.
- 67. Hall L, Colantonio A, Yoshida K. Barriers to nutrition as a health promotion practice for women with disabilities. International journal of rehabilitation research Internationale Zeitschrift fur Rehabilitationsforschung Revue internationale de recherches de readaptation.

- 2003;26(3):245-7. Epub 2003/09/23. doi: 10.1097/01.mrr.0000088450.78481.aa. PubMed PMID: 14501578.
- 68. Eisenberg Y, Vanderbom KA, Vasudevan V. Does the built environment moderate the relationship between having a disability and lower levels of physical activity? A systematic review. Preventive medicine. 2017;95s:S75-s84. Epub 2016/07/30. doi: 10.1016/j.ypmed.2016.07.019. PubMed PMID: 27471026.
- 69. Rimmer JH, Padalabalanarayanan S, Malone LA, Mehta T. Fitness facilities still lack accessibility for people with disabilities. Disability and health journal. 2016. Epub 2017/02/02. doi: 10.1016/j.dhjo.2016.12.011. PubMed PMID: 28143707.
- 70. Martin Ginis KA, Ma JK, Latimer-Cheung AE, Rimmer JH. A systematic review of review articles addressing factors related to physical activity participation among children and adults with physical disabilities. Health psychology review. 2016;10(4):478-94. Epub 2016/10/30. doi: 10.1080/17437199.2016.1198240. PubMed PMID: 27265062.
- 71. Donnelly JE, Goetz J, Gibson C, Sullivan DK, Lee R, Smith BK, Lambourne K, Mayo MS, Hunt S, Lee JH, Honas JJ, Washburn RA. Equivalent weight loss for weight management programs delivered by phone and clinic. Obesity (Silver Spring, Md). 2013;21(10):1951-9. Epub 2013/02/15. doi: 10.1002/oby.20334. PubMed PMID: 23408579; PMCID: Pmc4442605.
- 72. Donnelly JE, Pronk NP, Jacobsen DJ, Pronk SJ, Jakicic JM. Effects of a very-low-calorie diet and physical-training regimens on body composition and resting metabolic rate in obese females. American Journal of Clinical Nutrition. 1991;54:56-61.
- 73. Donnelly JE, Saunders RR, Saunders M, Washburn RA, Sullivan DK, Gibson CA, Ptomey LT, Goetz JR, Honas JJ, Betts JL, Rondon MR, Smith BK, Mayo MS. Weight management for individuals with intellectual and developmental disabilities: rationale and design for an 18 month randomized trial. Contemporary clinical trials. 2013;36(1):116-24. Epub 2013/07/03. doi: 10.1016/j.cct.2013.06.007. PubMed PMID: 23810939; PMCID: Pmc4180227.
- 74. Donnelly JE, Smith BK, Dunn L, Mayo MM, Jacobsen DJ, Stewart EE, Gibson CG, Sullivan D, K. Comparison of a phone vs clinic approach to achieve 10% weight loss. International Journal of Obesity. 2007;31:1270-6.
- 75. Donnelly JE, Sullivan DK, Smith BK, Jacobsen DJ, Washburn RA, Johnson SL, Hill JO, Mayo MS, Spaeth KR, Gibson C. Alteration of dietary fat intake to prevent weight gain: Jayhawk Observed Eating Trial. Obesity (Silver Spring, Md). 2008;16(1):107-12. Epub 2008/01/29. doi: 10.1038/oby.2007.33. PubMed PMID: 18223621.
- 76. Lambourne K, Washburn RA, Gibson C, Sullivan DK, Goetz J, Lee R, Smith BK, Mayo MS, Donnelly JE. Weight management by phone conference call: a comparison with a traditional face-to-face clinic. Rationale and design for a randomized equivalence trial. Contemporary clinical trials. 2012;33(5):1044-55. Epub 2012/06/06. doi: 10.1016/j.cct.2012.05.014. PubMed PMID: 22664647; PMCID: Pmc3408567.
- 77. Ptomey LT, Willis EA, Goetz JR, Lee J, Szabo-Reed AN, Sullivan DK, Donnelly JE. Portion-controlled meals provide increases in diet quality during weight loss and maintenance. Journal of human nutrition and dietetics: the official journal of the British Dietetic Association. 2015. Epub 2015/02/11. doi: 10.1111/jhn.12296. PubMed PMID: 25664818.
- 78. Ptomey LT, Sullivan DK, Lee J, Goetz JR, Gibson C, Donnelly JE. The use of technology for delivering a weight loss program for adolescents with intellectual and developmental disabilities. Journal of the Academy of Nutrition and Dietetics. 2015;115(1):112-8. Epub 2014/12/03. doi: 10.1016/j.jand.2014.08.031. PubMed PMID: 25441960.
- 79. LeCheminant JD, Gibson CA, Sullivan DK, Hall S, Washburn R, Vernon MC, Curry C, Stewart E, Westman EC, Donnelly JE. Comparison of a low carbohydrate and low fat diet for

- weight maintenance in overweight or obese adults enrolled in a clincial weight management program. Nutrition Journal. 2007;6(36).
- 80. LeCheminant JD, Jacobsen DJ, Hall MA, Donnelly JE. A comparison of meal replacements and medication in weight maintenance after weight loss. Journal of the American College of Nutrition. 2005;24:347-53.
- 81. Sullivan DK, Goetz JR, Gibson CA, Mayo MS, Washburn RA, Lee Y, Ptomey LT, Donnelly JE. A virtual reality intervention (second life) to improve weight maintenance: Rationale and design for an 18 month randomized trial. Contemporary clinical trials. 2015. Epub 2015/12/01. doi: 10.1016/j.cct.2015.11.019. PubMed PMID: 26616535.
- 82. Sullivan DK, Goetz JR, Gibson CA, Washburn RA, Smith BK, Lee J, Gerald S, Fincham T, Donnelly JE. Improving weight maintenance using virtual reality (Second Life). J Nutr Educ Behav. 2013;45(3):264-8. Epub 2013/04/30. doi: 10.1016/j.jneb.2012.10.007. PubMed PMID: 23622351.
- 83. Ptomey LT, Gibson CA, Lee J, Sullivan DK, Washburn RA, Gorczyca AM, Donnelly JE. Caregivers' effect on weight management in adults with intellectual and developmental disabilities. Disability and health journal. 2017. Epub 2017/02/22. doi: 10.1016/j.dhjo.2017.02.001. PubMed PMID: 28215627.
- 84. Willis EA, Szabo-Reed AN, Ptomey LT, Steger FL, Honas JJ, Al-Hihi EM, Lee R, Vansaghi L, Washburn RA, Donnelly JE. Distance learning strategies for weight management utilizing social media: A comparison of phone conference call versus social media platform. Rationale and design for a randomized study. Contemporary clinical trials. 2016;47:282-8. Epub 2016/02/18. doi: 10.1016/j.cct.2016.02.005. PubMed PMID: 26883282; PMCID: PMC4889333.
- 85. Froehlich-Grobe K, Aaronson LS, Washburn RA, Little TD, Lee J, Nary DE, Vansciver A, Nesbitt J, Norman SE. An exercise trial for wheelchair users: project workout on wheels. Contemporary clinical trials. 2012;33(2):351-63. Epub 2011/11/22. doi: 10.1016/j.cct.2011.10.014. PubMed PMID: 22101206; PMCID: Pmc3268824.
- 86. Nary DE, Froehlich-Grobe K, Aaronson L. Recruitment issues in a randomized controlled exercise trial targeting wheelchair users. Contemporary clinical trials. 2011;32(2):188-95. Epub 2010/11/03. doi: 10.1016/j.cct.2010.10.010. PubMed PMID: 21035565; PMCID: Pmc3034787.
- 87. Froehlich-Grobe K, Nary DE, Van Sciver A, Lee J, Little TD. Measuring height without a stadiometer: empirical investigation of four height estimates among wheelchair users. American journal of physical medicine & rehabilitation / Association of Academic Physiatrists. 2011;90(8):658-66. Epub 2011/06/18. doi: 10.1097/PHM.0b013e31821f6eb2. PubMed PMID: 21681063; PMCID: Pmc3148840.
- 88. Ptomey LT, Herrmann SD, Lee J, Sullivan DK, Rondon MF, Donnelly JE. Photo-assisted recall increases estimates of energy and macronutrient intake in adults with intellectual and developmental disabilities. Journal of the Academy of Nutrition and Dietetics. 2013;113(12):1704-9. Epub 2013/10/08. doi: 10.1016/j.jand.2013.07.029. PubMed PMID: 24095784; PMCID: Pmc3834035.
- 89. Saunders RP, Pate RR, Dowda M, Ward DS, Epping JN, Dishman RK. Assessing sustainability of Lifestyle Education for Activity Program (LEAP). Health education research. 2012;27(2):319-30. Epub 2011/12/14. doi: 10.1093/her/cyr111. PubMed PMID: 22156233; PMCID: PMC3303207.
- 90. Szabo-Reed AN, Lee J, Ptomey L, Willis E, Schubert M, Washburn R, Donnelly JE. Longitudinal Weight Loss Patterns and their Behavioral and Demographic Associations. Annals of behavioral medicine: a publication of the Society of Behavioral Medicine. 2016;50(1):147-56.

- Epub 2015/10/02. doi: 10.1007/s12160-015-9740-1. PubMed PMID: 26423446; PMCID: PMC4744131.
- 91. Yank V, Xiao L, Wilson SR, Stafford RS, Rosas LG, Ma J. Short-term weight loss patterns, baseline predictors, and longer-term follow-up within a randomized controlled trial. Obesity (Silver Spring, Md). 2014;22(1):45-51. Epub 2013/06/07. doi: 10.1002/oby.20510. PubMed PMID: 23740619; PMCID: Pmc3815705.
- 92. Nackers LM, Ross KM, Perri MG. The association between rate of initial weight loss and long-term success in obesity treatment: does slow and steady win the race? International journal of behavioral medicine. 2010;17(3):161-7. Epub 2010/05/06. doi: 10.1007/s12529-010-9092-y. PubMed PMID: 20443094; PMCID: Pmc3780395.
- 93. Hartmann-Boyce J, Johns DJ, Jebb SA, Aveyard P. Effect of behavioural techniques and delivery mode on effectiveness of weight management: systematic review, meta-analysis and meta-regression. Obesity reviews: an official journal of the International Association for the Study of Obesity. 2014;15(7):598-609. Epub 2014/03/19. doi: 10.1111/obr.12165. PubMed PMID: 24636238.
- 94. Hartmann-Boyce J, Johns DJ, Jebb SA, Summerbell C, Aveyard P. Behavioural weight management programmes for adults assessed by trials conducted in everyday contexts: systematic review and meta-analysis. Obesity reviews: an official journal of the International Association for the Study of Obesity. 2014;15(11):920-32. Epub 2014/08/13. doi: 10.1111/obr.12220. PubMed PMID: 25112559.
- 95. Nutrition AAoDa. How effective (in terms of client adherence and weight loss and maintenance) are meal replacements (liguid meals, meal bars, frozen prepackaged means)? 2011.
- 96. Lutes LD, Dinatale E, Goodrich DE, Ronis DL, Gillon L, Kirsh S, Richardson CR, Damschroder LJ. A randomized trial of a small changes approach for weight loss in veterans: design, rationale, and baseline characteristics of the ASPIRE-VA trial. Contemporary clinical trials. 2013;34(1):161-72. Epub 2012/10/09. doi: 10.1016/j.cct.2012.09.007. PubMed PMID: 23041618.
- 97. Damschroder LJ, Lutes LD, Kirsh S, Kim HM, Gillon L, Holleman RG, Goodrich DE, Lowery JC, Richardson CR. Small-changes obesity treatment among veterans: 12-month outcomes. American journal of preventive medicine. 2014;47(5):541-53. Epub 2014/09/14. doi: 10.1016/j.amepre.2014.06.016. PubMed PMID: 25217098.
- 98. Minniti A, Bissoli L, Di Francesco V, Fantin F, Mandragona R, Olivieri M, Fontana G, Rinaldi C, Bosello O, Zamboni M. Individual versus group therapy for obesity: comparison of dropout rate and treatment outcome. Eating and weight disorders: EWD. 2007;12(4):161-7. Epub 2008/01/30. PubMed PMID: 18227637.
- 99. Renjilian DA, Perri MG, Nezu AM, McKelvey WF, Shermer RL, Anton SD. Individual versus group therapy for obesity: effects of matching participants to their treatment preferences. Journal of consulting and clinical psychology. 2001;69(4):717-21. Epub 2001/09/12. PubMed PMID: 11550739.
- 100. Cresci B, Tesi F, La Ferlita T, Ricca V, Ravaldi C, Rotella CM, Mannucci E. Group versus individual cognitive-behavioral treatment for obesity: results after 36 months. Eating and weight disorders: EWD. 2007;12(4):147-53. Epub 2008/01/30. PubMed PMID: 18227635.
- 101. Lysandropoulos AP, Havrdova E. 'Hidden' factors influencing quality of life in patients with multiple sclerosis. European journal of neurology. 2015;22 Suppl 2:28-33. Epub 2015/09/17. doi: 10.1111/ene.12801. PubMed PMID: 26374511.

- 102. Russell D. Living arrangements, social integration, and loneliness in later life: the case of physical disability. Journal of health and social behavior. 2009;50(4):460-75. Epub 2010/01/27. PubMed PMID: 20099451.
- 103. Burke LE, Wang J, Sevick MA. Self-monitoring in weight loss: a systematic review of the literature. Journal of the American Dietetic Association. 2011;111(1):92-102. Epub 2010/12/28. doi: 10.1016/j.jada.2010.10.008. PubMed PMID: 21185970; PMCID: PMC3268700.
- 104. Semper HM, Povey R, Clark-Carter D. A systematic review of the effectiveness of smartphone applications that encourage dietary self-regulatory strategies for weight loss in overweight and obese adults. Obesity reviews: an official journal of the International Association for the Study of Obesity. 2016;17(9):895-906. Epub 2016/05/19. doi: 10.1111/obr.12428. PubMed PMID: 27192162.
- 105. Dale O, Hagen KB. Despite technical problems personal digital assistants outperform pen and paper when collecting patient diary data. Journal of clinical epidemiology. 2007;60(1):8-17. Epub 2006/12/13. doi: 10.1016/j.jclinepi.2006.04.005. PubMed PMID: 17161749.
- 106. Acharya SD, Elci OU, Sereika SM, Styn MA, Burke LE. Using a personal digital assistant for self-monitoring influences diet quality in comparison to a standard paper record among overweight/obese adults. Journal of the American Dietetic Association. 2011;111(4):583-8. Epub 2011/03/30. doi: 10.1016/j.jada.2011.01.009. PubMed PMID: 21443993; PMCID: PMC3406749.
- 107. Zheng Y, Burke LE, Danford CA, Ewing LJ, Terry MA, Sereika SM. Patterns of self-weighing behavior and weight change in a weight loss trial. International journal of obesity (2005). 2016;40(9):1392-6. Epub 2016/04/27. doi: 10.1038/ijo.2016.68. PubMed PMID: 27113642.
- 108. Zheng Y, Klem ML, Sereika SM, Danford CA, Ewing LJ, Burke LE. Self-weighing in weight management: A systematic literature review. Obesity (Silver Spring, Md). 2015;23(2):256-65. Epub 2014/12/19. doi: 10.1002/oby.20946. PubMed PMID: 25521523. 109. Zheng Y, Sereika SM, Ewing LJ, Danford CA, Terry MA, Burke LE. Association between Self-Weighing and Percent Weight Change: Mediation Effects of Adherence to Energy Intake and Expenditure Goals. Journal of the Academy of Nutrition and Dietetics. 2016;116(4):660-6. Epub 2016/01/05. doi: 10.1016/j.jand.2015.10.014. PubMed PMID: 26727241; PMCID: PMC4808617.
- 110. Szabo AN, Washburn RA, Sullivan DK, Honas JJ, Mayo MS, Goetz J, Lee J, Donnelly JE. The Midwest Exercise Trial for the Prevention of Weight Regain: MET POWeR. Contemporary clinical trials. 2013;36(2):470-8. Epub 2013/09/10. doi:
- 10.1016/j.cct.2013.08.011. PubMed PMID: 24012915; PMCID: PMC3844028.
- 111. Michie S, Abraham C, Whittington C, McAteer J, Gupta S. Effective techniques in healthy eating and physical activity interventions: a meta-regression. Health psychology: official journal of the Division of Health Psychology, American Psychological Association. 2009;28(6):690-701. Epub 2009/11/18. doi: 10.1037/a0016136. PubMed PMID: 19916637.
- 112. Golden SD, Earp JA. Social ecological approaches to individuals and their contexts: twenty years of health education & behavior health promotion interventions. Health education & behavior: the official publication of the Society for Public Health Education. 2012;39(3):364-72. Epub 2012/01/24. doi: 10.1177/1090198111418634. PubMed PMID: 22267868.
- 113. (NCHS) NCfHS. Physical Function items of the National Health and Nutrition Examination Survey1999-2000.
- 114. Wilt TJ, Carlson KF, Goldish GD, MacDonald R, Niewoehner C, Rutks I, Shamliyan T, Tacklind J, Taylor BC, Kane RL. Carbohydrate and lipid disorders and relevant considerations in

- persons with spinal cord injury. Evidence report/technology assessment. 2008(163):1-95. Epub 2008/05/07. PubMed PMID: 18457480.
- 115. Laughton GE, Buchholz AC, Martin Ginis KA, Goy RE. Lowering body mass index cutoffs better identifies obese persons with spinal cord injury. Spinal cord. 2009;47(10):757-62. Epub 2009/04/08. doi: 10.1038/sc.2009.33. PubMed PMID: 19350042.
- 116. Ravensbergen HR, Lear SA, Claydon VE. Waist circumference is the best index for obesity-related cardiovascular disease risk in individuals with spinal cord injury. Journal of neurotrauma. 2014;31(3):292-300. Epub 2013/09/28. doi: 10.1089/neu.2013.3042. PubMed PMID: 24070685; PMCID: Pmc3904532.
- 117. Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addictive behaviors. 1982;7(1):47-55. Epub 1982/01/01. PubMed PMID: 7080884.
- 118. Garner DM, Olmsted MP, Bohr Y, Garfinkel PE. The eating attitudes test: psychometric features and clinical correlates. Psychological medicine. 1982;12(4):871-8. Epub 1982/11/01. PubMed PMID: 6961471.
- 119. Grossi E, Dalle Grave R, Mannucci E, Molinari E, Compare A, Cuzzolaro M, Marchesini G. Complexity of attrition in the treatment of obesity: clues from a structured telephone interview. International Journal of Obesity. 2006;30(7):1132.
- 120. Wadden TA, Letizia KA. Predictors of attrition and weight loss in patients treated by moderate and severe caloric restriction 1992.
- 121. Library AAoDaNEA. Practice Guidelines for Nutrition Care for Patients with Spinal Cord Injury. <a href="http://adaevidencealibrary.com">http://adaevidencealibrary.com</a>: 2009.
- 122. Ditschuneit HH, Flechtner-Mors M. Value of structured meals for weight management: risk factors and long-term weight maintenance. Obesity research. 2001;9 Suppl 4:284s-9s. Epub 2001/11/15. doi: 10.1038/oby.2001.132. PubMed PMID: 11707555.
- 123. Bauman WA, Spungen AM, Wang J, Pierson RN, Jr. The relationship between energy expenditure and lean tissue in monozygotic twins discordant for spinal cord injury. Journal of rehabilitation research and development. 2004;41(1):1-8. Epub 2004/07/27. PubMed PMID: 15273892.
- 124. Buchholz AC, McGillivray CF, Pencharz PB. Differences in resting metabolic rate between paraplegic and able-bodied subjects are explained by differences in body composition. The American journal of clinical nutrition. 2003;77(2):371-8. Epub 2003/01/24. PubMed PMID: 12540396.
- 125. Feasel S, Groah SL. The impact of diet on cardiovascular disease risk in individuals wih spinal cord injury. Topics in Spinal Cord Injury Relabilitation. 2009;14(3):58-68.
- 126. Khalil RE, Gorgey AS, Janisko M, Dolbow DR, Moore JR, Gater DR. The role of nutrition in health status after spinal cord injury. Aging and disease. 2013;4(1):14-22. Epub 2013/02/21. PubMed PMID: 23423356; PMCID: Pmc3570137.
- 127. Cox SA, Weiss SM, Posuniak EA, Worthington P, Prioleau M, Heffley G. Energy expenditure after spinal cord injury: an evaluation of stable rehabilitating patients. The Journal of trauma. 1985;25(5):419-23. Epub 1985/05/01. PubMed PMID: 3999162.
- 128. Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. American Journal of Clinical Nutrition. 1990;51:241-7.
- 129. Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: Updated recommendation for

- adults from the American College of Sports Medicine and the American Heart Association. Medicine & Science in Sports & Exercise. 2007;39(8):1423-34.
- 130. Services USDoHaH. Physical activity guidelines advisory committee report to the Secretary of Health and Human Services2008.
- 131. Ginis KA, Arbour-Nicitopoulos KP, Latimer AE, Buchholz AC, Bray SR, Craven BC, Hayes KC, Hicks AL, McColl MA, Potter PJ, Smith K, Wolfe DL. Leisure time physical activity in a population-based sample of people with spinal cord injury part II: activity types, intensities, and durations. Archives of physical medicine and rehabilitation. 2010;91(5):729-33. Epub 2010/05/04. doi: 10.1016/j.apmr.2009.12.028. PubMed PMID: 20434610.
- 132. Wilroy J, Knowlden A. Systematic review of theory-based interventions aimed at increasing physical ativity in individuals with spinal cord injury. American Journal of Health Education. 2016;47(3):163-74.
- 133. Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Medicine & Science in Sports & Exercise. 2009;41(2):459-71.
- 134. Kressler J, Cowan RE, Bigford GE, Nash MS. Reducing cardiometabolic disease in spinal cord injury. Physical medicine and rehabilitation clinics of North America. 2014;25(3):573-604, viii. Epub 2014/07/30. doi: 10.1016/j.pmr.2014.04.006. PubMed PMID: 25064789.
- 135. Shuval K, Finley CE, Barlow CE, Nguyen BT, Njike VY, Pettee Gabriel K. Independent and joint effects of sedentary time and cardiorespiratory fitness on all-cause mortality: the Cooper Center Longitudinal Study. BMJ open. 2015;5(10):e008956. Epub 2015/11/04. doi: 10.1136/bmjopen-2015-008956. PubMed PMID: 26525421; PMCID: Pmc4636648.
- 136. Pulsford RM, Stamatakis E, Britton AR, Brunner EJ, Hillsdon MM. Sitting behavior and obesity: evidence from the Whitehall II study. American journal of preventive medicine. 2013;44(2):132-8. doi: 10.1016/j.amepre.2012.10.009. PubMed PMID: 23332328; PMCID: 3550520.
- 137. Manns PJ, Dunstan DW, Owen N, Healy GN. Addressing the nonexercise part of the activity continuum: a more realistic and achievable approach to activity programming for adults with mobility disability? Physical therapy. 2012;92(4):614-25. Epub 2011/12/14. doi: 10.2522/ptj.20110284. PubMed PMID: 22156025.
- 138. Bai Y, Welk GJ, Nam YH, Lee JA, Lee JM, Kim Y, Meier NF, Dixon PM. Comparison of Consumer and Research Monitors under Semistructured Settings. Medicine and science in sports and exercise. 2016;48(1):151-8. Epub 2015/07/15. doi:
- 10.1249/mss.0000000000000727. PubMed PMID: 26154336.
- 139. Nelson MB, Kaminsky LA, Dickin DC, Montoye AH. Validity of Consumer-Based Physical Activity Monitors for Specific Activity Types. Medicine and science in sports and exercise. 2016;48(8):1619-28. Epub 2016/03/26. doi: 10.1249/mss.0000000000000933. PubMed PMID: 27015387.
- 140. Nary D. Accessible Scales Support Health for Wheelchair Users 2013.
- 141. Graham CL, Mann JR. Accessibility of primary care physician practice sites in South Carolina for people with disabilities. Disability and health journal. 2008;1(4):209-14. Epub 2008/10/01. doi: 10.1016/j.dhjo.2008.06.001. PubMed PMID: 21122731.
- 142. Mudrick NR, Breslin ML, Liang M, Yee S. Physical accessibility in primary health care settings: results from California on-site reviews. Disability and health journal. 2012;5(3):159-67. Epub 2012/06/26. doi: 10.1016/j.dhjo.2012.02.002. PubMed PMID: 22726856.

- 143. Pharr J. Accessible medical equipment for patients with disabilities in primary care clinics: why is it lacking? Disability and health journal. 2013;6(2):124-32. Epub 2013/03/20. doi: 10.1016/j.dhjo.2012.11.002. PubMed PMID: 23507163.
- 144. Lohman TG, Roche AF, Martorell R. Anthropometric standardization reference manual. Champaign,III: Human Kinetics Books; 1988 1988.
- 145. Centers fDCa, Prevention. National Health and Nutrition Survey (NHANES):Health Tech/Blood Pressure Procedures Manual. Atlanta, GA: Center for Disease Control and Prevention; 2009.
- 146. WHO Guidelines on drawing blood: best practices in phlebotomy. Geneva, Switzerland: WHO Document Production Services; 2010.
- 147. Ware JE, Jr., Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Medical care. 1992;30(6):473-83. Epub 1992/06/11. PubMed PMID: 1593914.
- 148. Ware JE, Snow KK, Kosinski M, Gandek B. SF-36 health survey: manual and interpretation guide. In: Institute TH, editor. Boston, MA1993.
- 149. Froehlich-Grobe K, Andresen EM, Caburnay C, White GW. Measuring health-related quality of life for persons with mobility impairments: an enabled version of the short-form 36 (SF-36E). Quality of life research: an international journal of quality of life aspects of treatment, care and rehabilitation. 2008;17(5):751-70. Epub 2008/04/23. doi: 10.1007/s11136-008-9342-5. PubMed PMID: 18427950.
- 150. Drummond MF, Sculpher MJ, Torrance GW. Methods for Economic Evlauation of Health Care Programs. Oxford, UK: Oxford University Press; 2005.
- 151. Narbro K, Sjostrom L. Willingness to pay for obesity treatment. International journal of technology assessment in health care. 2000;16(1):50-9. Epub 2000/05/18. PubMed PMID: 10815353.
- 152. Sloan FA. Valuing Health Care: Costs, Benefits, and Effectiveness of Pharmaceuticals and other Medical Technologies. Cambridge, UK: Cambridge University Press; 1996.
- 153. Lee RH, Bott MJ, Forbes S, Redford L, Swagerty DL, Taunton RL. Process-based costing. Journal of nursing care quality. 2003;18(4):259-66. Epub 2003/10/15. PubMed PMID: 14556582.
- 154. Russell LB, Gold MR, Siegel JE, Daniels N, Weinstein MC. The role of cost-effectiveness analysis in health and medicine. Panel on Cost-Effectiveness in Health and Medicine. Jama. 1996;276(14):1172-7. Epub 1996/10/09. PubMed PMID: 8827972.
- 155. Frew E, Wolstenholme JL, Atkin W, Whynes DK. Estimating time and travel costs incurred in clinic based screening: flexible sigmoidoscopy screening for colorectal cancer. Journal of medical screening. 1999;6(3):119-23. Epub 1999/11/26. PubMed PMID: 10572841.
- 156. Yabroff KR, Warren JL, Knopf K, Davis WW, Brown ML. Estimating patient time costs associated with colorectal cancer care. Medical care. 2005;43(7):640-8. Epub 2005/06/23. PubMed PMID: 15970778.
- 157. Reuben DB, Wong RC, Walsh KE, Hays RD. Feasibility and accuracy of a postcard diary system for tracking healthcare utilization of community-dwelling older persons. Journal of the American Geriatrics Society. 1995;43(5):550-2. Epub 1995/05/01. PubMed PMID: 7730540.
- 158. Ptomey LT, Willis EA, Goetz JR, Lee J, Sullivan DK, Donnelly JE. Digital photography improves estimates of dietary intake in adolescents with intellectual and developmental disabilities. Disability and health journal. 2015;8(1):146-50. Epub 2014/10/05. doi: 10.1016/j.dhjo.2014.08.011. PubMed PMID: 25281035.

- 159. Humphries K, Traci MA, Seekins T. Food on file: Pilot test of an innovative method for recording food intake of adults with intellectual disabilities living in the community. Journal of Applied Research in Intellectual Disabilities. 2008;21(2):126-73.
- 160. Ptomey LT, Willis EA, Honas JJ, Mayo MS, Washburn RA, Herrmann SD, Sullivan DK, Donnelly JE. Validity of energy intake estimated by digital photography plus recall in overweight and obese young adults. Journal of the Academy of Nutrition and Dietetics. 2015;115(9):1392-9.
- 161. Rimmer JH, Riley BB, Rubin SS. A new measure for assessing the physical activity behaviors of persons with disabilities and chronic health conditions: the Physical Activity and Disability Survey. American journal of health promotion: AJHP. 2001;16(1):34-42. Epub 2001/09/29. PubMed PMID: 11575054.
- 162. Rimmer JH, Rauworth A, Wang E, Heckerling PS, Gerber BS. A randomized controlled trial to increase physical activity and reduce obesity in a predominantly African American group of women with mobility disabilities and severe obesity. Preventive medicine. 2009;48(5):473-9. Epub 2009/05/22. PubMed PMID: 19459233.
- 163. Clark M, Abrams DB, Niaura RS. Self-efficacy in weight management. Journal of consulting and clinical psychology. 1991;59:739-44.
- 164. Grandy S, Hashemi M, Langkilde AM, Parikh S, Sjostrom CD. Changes in weight loss-related quality of life among type 2 diabetes mellitus patients treated with dapagliflozin. Diabetes, obesity & metabolism. 2014;16(7):645-50. Epub 2014/01/22. doi: 10.1111/dom.12263. PubMed PMID: 24443876.
- 165. Fontaine KR, Cheskin LJ. Self-efficacy, attendance, and weight loss in obesity treatment. Addictive behaviors. 1997;22(4):567-70. Epub 1997/07/01. PubMed PMID: 9290865. 166. Kroll T, Kehn M, Ho PS, Groah S. The SCI Exercise Self-Efficacy Scale (ESES):
- development and psychometric properties. The international journal of behavioral nutrition and physical activity. 2007;4:34. Epub 2007/09/01. doi: 10.1186/1479-5868-4-34. PubMed PMID: 17760999: PMCID: Pmc2034591.
- 167. Becker H, Stuifbergen AK, Sands D. Development of a scale to measure barriers to health promotion activities among persons with disabilities. American journal of health promotion: AJHP. 1991;5(6):449-54. Epub 1991/06/08. PubMed PMID: 10171668.
- 168. Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. Journal of psychosomatic research. 1985;29(1):71-83. Epub 1985/01/01. PubMed PMID: 3981480.
- 169. Cappelleri JC, Bushmakin AG, Gerber RA, Leidy NK, Sexton CC, Lowe MR, Karlsson J. Psychometric analysis of the Three-Factor Eating Questionnaire-R21: results from a large diverse sample of obese and non-obese participants. International journal of obesity (2005). 2009;33(6):611-20. Epub 2009/04/29. doi: 10.1038/ijo.2009.74. PubMed PMID: 19399021.
- 170. Angle S, Engblom J, Eriksson T, Kautiainen S, Saha MT, Lindfors P, Lehtinen M, Rimpela A. Three factor eating questionnaire-R18 as a measure of cognitive restraint, uncontrolled eating and emotional eating in a sample of young Finnish females. The international journal of behavioral nutrition and physical activity. 2009;6:41. Epub 2009/07/21. doi: 10.1186/1479-5868-6-41. PubMed PMID: 19615047; PMCID: Pmc2720907.
- 171. Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Preventive medicine. 1987;16(6):825-36. Epub 1987/11/01. PubMed PMID: 3432232.
- 172. Buysse DJ, Reynolds CF, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry research. 1989;28(2):193-213.

- 173. Lobentanz I, Asenbaum S, Vass K, Sauter C, Klösch G, Kollegger H, Kristoferitsch W, Zeitlhofer J. Factors influencing quality of life in multiple sclerosis patients: disability, depressive mood, fatigue and sleep quality. Acta Neurologica Scandinavica. 2004;110(1):6-13.
- 174. Chien M-Y, Chen H-C. Poor sleep quality is independently associated with physical disability in older adults. Journal of clinical sleep medicine: JCSM: official publication of the American Academy of Sleep Medicine. 2015;11(3):225.
- 175. Domecq JP, Prutsky G, Leppin A, Sonbol MB, Altayar O, Undavalli C, Wang Z, Elraiyah T, Brito JP, Mauck KF, Lababidi MH, Prokop LJ, Asi N, Wei J, Fidahussein S, Montori VM, Murad MH. Clinical review: Drugs commonly associated with weight change: a systematic review and meta-analysis. The Journal of clinical endocrinology and metabolism.
- 2015;100(2):363-70. Epub 2015/01/16. doi: 10.1210/jc.2014-3421. PubMed PMID: 25590213.
- 176. Ditschuneit HH, Flechtner-Mors M, Johnson TD, Adler G. Metabolic and weight-loss effects of a long-term dietary intervention in obese patients. The American journal of clinical nutrition. 1999;69(2):198-204. Epub 1999/02/16. PubMed PMID: 9989680.
- 177. Flechtner-Mors M, Ditschuneit HH, Johnson TD, Suchard MA, Adler G. Metabolic and weight loss effects of long-term dietary intervention in obese patients: four-year results. Obesity research. 2000;8(5):399-402. Epub 2000/09/01. doi: 10.1038/oby.2000.48. PubMed PMID: 10968732.
- 178. Lalonde L, Gray-Donald K, Lowensteyn I, Marchand S, Dorais M, Michaels G, Llewellyn-Thomas HA, O'Connor A, Grover SA. Comparing the benefits of diet and exercise in the treatment of dyslipidemia. Preventive medicine. 2002;35(1):16-24. Epub 2002/06/25. PubMed PMID: 12079437.
- 179. Stevens J, Truesdale KP, McClain JE, Cai J. The definition of weight maintenance. International journal of obesity (2005). 2006;30(3):391-9. Epub 2005/11/23. doi: 10.1038/sj.ijo.0803175. PubMed PMID: 16302013.
- 180. Truesdale KP, Stevens J, Cai J. The effect of weight history on glucose and lipids: the Atherosclerosis Risk in Communities Study. American journal of epidemiology. 2005;161(12):1133-43. Epub 2005/06/07. doi: 10.1093/aje/kwi151. PubMed PMID: 15937022;

PMCID: PMC3234677.

181. Saunders RR, Saunders MD, Donnelly JE, Smith BK, Sullivan DK, Guilford B, Rondon MF. Evaluation of an approach to weight loss in adults with intellectual or developmental disabilities. Intellectual and developmental disabilities. 2011;49(2):103-12. Epub 2011/03/31. doi: 10.1352/1934-9556-49.2.103. PubMed PMID: 21446873.